CLINICAL TRIAL: NCT01374776
Title: Effect Of Intravenous Iron Versus Placebo On Muscle Oxidative Capacity And Physical Performance In Non Anemic Premenopausal Women With Low Ferritin Levels
Brief Title: Effect Of Intravenous Iron Versus Placebo On Muscle Oxidative Capacity And Physical Performance in Premenopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Version number 2 fro
Record Dates: First submitted 2011-06-15; First posted 2011-06-16 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Non Anemic Patients With Iron Deficiency (Low Ferritin Value)

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (1):
- intravenous iron carboxymaltose (Experimental): intravenous iron carboxymaltose infusion
  Interventions: Drug: intravenous iron carboxymaltose

INTERVENTIONS:
Drug: intravenous iron carboxymaltose — The patients will be randomized to one of the 2 treatment groups (12 patients in each group): Group I: intravenous iron carboxymaltose; Group II: intravenous placebo. Group I (intravenous iron): Ferinject will be applied via a short infusion. Patients will receive 15mg/kg of iron as iron carboxymaltose Ferinject® in 250 ml 0.9% NaCl intravenously (time of infusion 20 mins), in a single dose. The maximum dose is limited to 1000mg iron. Group II (intravenous placebo): Intravenous placebo (250 ml 0.9 % NaCl will be administrated in the same manner and time schedule than group I.

SUMMARY:
Effect of intravenous iron substitution (iron carboxymaltose (Ferinject®), total dose 15 mg/ kg (maximal dose: 1000mg) in 250 ml 0.9 % NaCl; intravenous infusion in 20 min)in non-anemic premenopausal women with iron deficiency on

Primary objective:

- Mitochondrial capacity (Phosphocreatine Recovery rate assessed by 31P-MR-spectroscopy of the lower leg muscle)

Secondary objectives:

* Maximal oxygen uptake during a graded cycling exercise test and time to exhaustion at submaximal power during a constant-load cycling exercise test
* Plantarflexor muscle fatiguability as assessed by isokinetic dynamometry
* Trial with medicinal product

ELIGIBILITY:
Inclusion criteria: INCLUSION CRITERIA

* Healthy female subjects, Age > 18 years, premenopausal, regularly menstruating
* BMI 18-25 kg/m2.
* Serum ferritin level < 15ug/ml
* Recreationally active with = 1.5 h/w structured activity
* Adequate contraception during the study period
* Informed consent

Exclusion criteria: EXCLUSION CRITERIA

* Anemia with Hb level < 120 g/l
* Known hypersensitivity to iron carboxymaltose, iron sucrose or iron sulfate
* Intake of iron preparations (also multivitamins containing iron) during the last 8 weeks before the start of the trial protocol
* Pregnancy or lactation
* Any cardiovascular or pulmonary disease
* Any orthopaedic or rheumatologic disease which affects exercise performance
* Presence of muscle disease
* Acute or chronic infection/inflammation or malignancy
* Known mental disorders (e.g. depression)
* Intake of concurrent medication, except oral contraceptives
* CRP > 10 mg/l
* TSH out of normal range
* Elevated CK (> 167 U/l)
* Any concurrent medical condition(s) that, in the view of the investigator, would prevent compliance or participation or jeopardize the health of the patients.
* Participation in any other therapeutic trial within the previous month

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Mitochondrial capacity (Phosphocreatine Recovery rate assessed by 31P-MR-spectroscopy of the lower leg muscle) | one year

CONTACTS AND LOCATIONS:
Overall Officials: Pierre-Alexandre Krayenbuehl, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Clinic and Policlinic of Internal Medicine, Zurich, Canton of Zurich, Switzerland